CLINICAL TRIAL: NCT02282956
Title: Monocentric, Non-blinded, Prospective Randomized Parallel Group Phase IV Clinical Study to Evaluate the Efficacy of Ultrasound Guided Single Shot Block of Nervus Tibialis Posterior for Postoperative Pain Relief After Hallux Valgus Surgery.
Brief Title: Ultrasound Guided Single Shot Block of Posterior Tibial Nerve for Postoperative Pain Relief After Hallux Valgus Surgery
Acronym: Hallux
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr.med. Sabine Schoenfeld (Other)
Responsible Party: Sponsor-Investigator, Dr.med. Sabine Schoenfeld, senior consultant for anesthesia, Spitalregion Rheintal, Werdenberg, Sarganserland
Organization: Spitalregion Rheintal, Werdenberg, Sarganserland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 13/126
Record Dates: First submitted 2014-10-27; First posted 2014-11-05 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus | interventions — Morphine; Droperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): single shot, posterior tibial nerve block with 5 ml of Ropivacaine 0,75% before surgery postoperative PCA pump with morphine and droperidol (DHBP®) for the next 24 hours.
  Interventions: Drug: Ropivacaine 0,75%; Procedure: posterior tibial nerve block; Drug: morphine and droperidol
- controll Group (Other): After surgery: standard analgesic treatment by PCA (patient controlled analgesia) pumps with morphine and Droperidol (DHBP®) for the next 24 hours.
  Interventions: Drug: morphine and droperidol

INTERVENTIONS:
Drug: Ropivacaine 0,75% — Ropivacaine injection
  Other Names: Naropin 0,75%
  Arms: study group
Procedure: posterior tibial nerve block — ultrasound guided posterior tibal nerve block
  Arms: study group
Drug: morphine and droperidol — i.v PCA
  Other Names: DHBP

SUMMARY:
Hallux surgery is known to be extremely painful. Standard pain therapy is treatment with NSAID and opioid painkillers. Patients are frequently not-satisfied with this. Some institutions use a nerve block (single shot or catheter technic) of the ischiadic nerve. But this procedure is invasive, has a potential risk of nerve lesion, and is not accepted by all surgeons. A single shot nerve block of the posterior tibial nerve is less invasive and could be superior compared to standard pain treatment. A great variability of nerve supply of the foot is well described. There are some hints that the posterior tibial nerve supplies the first metatarsal bone and the first metatarsal joint. A nerve block could reduce postoperative pain in hallux surgery. To assess the effectiveness of this investigated measure, the requested morphine dose of a PCA pump will be used to verify the effectiveness of the tibial nerve block.

DETAILED DESCRIPTION:
The overall purpose is to evaluate the effectiveness of tibial nerve block for postoperative pain relief after hallux surgery. The primary objective is to assess the morphine requirement in the first 24 hours after surgery. Secondary objectives are maximum pain scores and sleeping quality in the postoperative period. Patient's satisfaction with the pain therapy and approximately nerve block duration will be asked in the final interview.

Primary study endpoint is a 50% reduction of morphine requirement with a 60% standard deviation within 24 hours after surgery. Power is 80%, the level of significance is set at 5% (p < 0,05).

Secondary endpoints are sleeping quality and maximum pain scores (maximum VAS) measured by means of postoperative questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Elective Hallux valgus surgery ("Magerl" operation technique)

Exclusion Criteria:

* Patient refusal, pregnancy
* Regular medication with opioids
* Drug abuse
* Contraindication for regional anesthesia
* Known allergy against one of the study drugs
* Polyneuropathia, or any other neurodegenerative disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
morphine requirement | 24 hours
  a 50% reduction of morphine requirement with a 60% standard deviation within 24 hours after surgery. Power is 80%, the level of significance is set at 5% (p < 0,05).

SECONDARY OUTCOMES:
sleeping quality | 24 hours
  sleeping quality in the first postoperative night, questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Schoenfeld, MD, Principal Investigator — 9472 Grabs, Spitalstrasse 44, switzerland
Locations (1):
- Spital Grabs, Grabs, Switzerland

REFERENCES:
- [Background] Unlu RE, Orbay H, Kerem M, Esmer AF, Tuccar E, Sensoz O. Innervation of three weight-bearing areas of the foot: an anatomic study and clinical implications. J Plast Reconstr Aesthet Surg. 2008;61(5):557-61. doi: 10.1016/j.bjps.2007.02.007. Epub 2007 Apr 2. PMID 17400530
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed